CLINICAL TRIAL: NCT01009983
Title: A Phase II Clinical Trial of Weekly Paclitaxel and Carboplatin in Combination With Panitumumab in Metastatic Breast Cancer Patients With Triple Negative Disease
Brief Title: Paclitaxel, Carboplatin, and Panitumumab in Treating Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00010510; NCI-2009-01257 (Other: CTRP); CCCWFU74108 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
Keywords: triple-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Panitumumab; Paclitaxel; Taxes; Carboplatin; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients receive paclitaxel IV and carboplatin IV on days 1, 8, and 15. Patients also receive panitumumab IV on days 1 and 15.
  Interventions: Biological: panitumumab; Drug: paclitaxel; Drug: carboplatin; Procedure: laboratory biomarker analysis; Procedure: immunohistochemistry staining method

INTERVENTIONS:
Biological: panitumumab — Given IV
  Other Names: ABX-EGF; clone E7.6.3; MOAB ABX-EGF; monoclonal antibody ABX-EGF; Vectibix
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin; Paraplatine
Procedure: laboratory biomarker analysis — Correlative study
Procedure: immunohistochemistry staining method — Correlative study
  Other Names: immunohistochemistry

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Other find tumor cells and help kill them or carry tumor-killing substances to them. Giving panitumumab together with paclitaxel and carboplatin may be a better way to block tumor growth.

PURPOSE: This phase II trial is studying the side effects and how well paclitaxel and carboplatin together with panitumumab works in treating patients with metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the response rate to the combination of carboplatin, paclitaxel and panitumumab in women with ER-, PR- and Her-2 negative metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To determine the tolerability and toxicities of the combination of paclitaxel, carboplatin and panitumumab.

II. To determine the markers that co-occur with EGFR expression in the triple negative breast cancer.

III. To assess the association between tumor biomarkers and clinical outcomes (response and survival).

IV. To examine the effect this regimen has on time to progression and survival.

OUTLINE:

Patients receive paclitaxel IV and carboplatin IV on days 1, 8, and 15. Patients also receive panitumumab IV on days 1 and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion

* Pathologically confirmed invasive breast cancer with ER < 10%, PR < 10%, by IHC, HER2 1+ or 0 or FISH negative
* Measurable (>= 1 cm) or assessable disease detectable by imagining or physical exam
* Patients with bone only disease have measurable lesions on x-ray, MRI, or CT scan
* Only one or no prior therapy for metastatic or recurrent breast cancer is allowed
* Prior chemotherapy or radiation therapy is permitted but at least 2 weeks should elapse prior to study enrollment
* Prior therapy with bevacizumab is permitted but at least 2 weeks should elapse prior to study enrollment
* Prior therapy with bevacizumab is permitted but at least 28 days should elapse from the last bevacizumab treatment prior to study enrollment
* ECOG PS or 0-1
* Signed protocol specific informed consent prior to registration
* Life expectancy greater than 3 months
* Please contact study investigator and/or consult the protocol document for specific laboratory criteria
* Tissue block available from primary breast cancer
* Premenopausal women must have a negative serum or urine pregnancy test prior to starting on study treatment (post-menopausal is defined as > 6 months of amenorrhea prior hysterectomy)

Exclusion

* More than or equal to 2 prior regimens for metastatic breast cancer
* Leptomeningeal disease
* Brain metastasis except for a solitary lesion that was resected or treated with gamma knife with no residual disease on CT or MRI or received whole brain RT and f/u MRI was normal with no residual neurologic deficit
* History of interstitial lung disease (ie pneumonitis, pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest computerized tomography (CT) scan
* History of irreversible neuropathy
* Another malignancy other than carcinoma in situ of the cervix or skin cancer
* Active uncontrolled bacterial viral or fungal infection
* Active pregnancy or breast feeding
* Patients with pre-existing neuropathy >= grade 2
* History of myocardial infarction, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Patients with previous history of CTCAE grade >= 3 hypersensitivity to paclitaxel or Cremophor EL are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi D Klepin, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started | 14
Completed | 13
Not Completed | 1
Not completed — necessary scans not completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Activity as Assessed by Objective Tumor Response According to RECIST Criteria
Description: Complete or Partial response as defined by reduction in tumor size according to RECIST (Response Evaluation Criteria In Solid Tumors) rules.
Time Frame: every 28 days for a minimum of 84 days
Measure: Number; unit: participants
Arm/Group | Arm 1
Number analyzed (Participants) | 13
participants | 6

2. Secondary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Approximately 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 14
months | 5.3 [2.2 to 5.8]

3. Secondary Outcome: Survival
Time Frame: Approximately 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 14
months | 6.8 [3.1 to NA] — Due to calculation of confidence interval, the upper bound is not estimated because not enough of the sample had an event.

4. Secondary Outcome: Expression of EGFR and Other Protein Markers
Time Frame: baseline
Population: Test not completed as specified in protocol that will only be completed if a full sample was accrued.
Arm/Group | Arm 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=14)
Low WBC (Investigations) | 4 (4)
low Platelets (Investigations) | 1 (1)
Low Hemoglobin (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Alkaline phosphatase (Investigations) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Neuropathy: sensory (Cardiac disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Low ANC (Investigations) | 9 (9)
hyperglycemia (Investigations) | 2 (2)
hypoglycemia (Investigations) | 1 (1)
hypocalcemia (Investigations) | 2 (2)
hypomagnesemia (Investigations) | 2 (2)
hypokalemia (Investigations) | 1 (1)
hypoalbuminemia (Investigations) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
serum glutamic oxaloacetic transaminase (Investigations) | 1 (1)
Dehydration (General disorders) | 1 (1)
Pruritus/itching (General disorders) | 1 (1)
Pain: Breast (General disorders) | 1 (1)
Lymphopenia (Investigations) | 5 (5)
Pain: Extremity-limb (General disorders) | 1 (1)
Urinary with low grade neutropenia (Infections and infestations) | 1 (1)
blurred vision (Eye disorders) | 1 (1)
Death not associated with CTCAE term: Disease progression NOS (General disorders) | 1 (1)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 2 (2)
Hemorrhage, GI: Upper GI (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=14)
Low WBC (Investigations) | 7 (7)
low Platelets (Investigations) | 10 (10)
Low Hemoglobin (Investigations) | 12 (12)
Nausea (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Anorexia (General disorders) | 2 (2)
Alkaline phosphatase (Investigations) | 8 (8)
Creatinine (Investigations) | 1 (1)
Proteinuria (Investigations) | 3 (3)
Hair loss (General disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hypertension (General disorders) | 2 (2)
Hypotension (Cardiac disorders) | 5 (5)
Neuropathy: sensory (Cardiac disorders) | 8 (8)
Neuropathy: motor (Nervous system disorders) | 2 (2)
Low ANC (Investigations) | 5 (5)
Pain (General disorders) | 3 (3)
Dizziness (General disorders) | 4 (4)
Taste alteration (General disorders) | 1 (1)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 4 (4)
Rigors/chills (General disorders) | 1 (1)
Fatigue (General disorders) | 8 (8)
Weight loss (General disorders) | 3 (3)
hyperglycemia (Investigations) | 9 (9)
hypocalcemia (Investigations) | 5 (5)
hypomagnesemia (Investigations) | 11 (11)
hyponatremia (Investigations) | 3 (3)
hypokalemia (Investigations) | 9 (9)
Hot flashes/flushes (General disorders) | 1 (1)
Bicarbonate serum-low (Investigations) | 1 (1)
hypoalbuminemia (Investigations) | 6 (6)
hyperbilirubinemia (Investigations) | 4 (4)
serum glutamic pyruvic transaminase (Investigations) | 6 (6)
hypophosphatemia (Investigations) | 2 (2)
Constipation (Gastrointestinal disorders) | 8 (8)
Pain: Head/headache (General disorders) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
serum glutamic oxaloacetic transaminase (Investigations) | 4 (4)
hypermagnesemia (Investigations) | 1 (1)
Ocular/Visual - Other (Eye disorders) | 1 (1)
Fever without neutropenia (General disorders) | 4 (4)
Urinary frequency/urgency (General disorders) | 1 (1)
Infection - Other (Infections and infestations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema: limb (Vascular disorders) | 1 (1)
Speech impairment (General disorders) | 1 (1)
Dehydration (General disorders) | 2 (2)
Pruritus/itching (General disorders) | 1 (1)
Anxiety (General disorders) | 2 (2)
Depression (General disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (4)
Pain: Abdomen (General disorders) | 3 (3)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 7 (7)
Partial Thromboplastin Time (Investigations) | 1 (1)
Pain: Joint (General disorders) | 1 (1)
Ataxia (General disorders) | 1 (1)
Pain: Back (General disorders) | 3 (3)
Pain: Bone (General disorders) | 1 (1)
Pain: Breast (General disorders) | 1 (1)
Pain: Chest/thorax (General disorders) | 1 (1)
Pain: Chest wall (General disorders) | 1 (1)
Wound complication, non-infectious (General disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Hemorrhage respiratory (Vascular disorders) | 1 (1)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Extremity-lower (gait/walking) (General disorders) | 1 (1)
Glomerular filtration rate (Investigations) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Voice changes (General disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (3)
Lymphopenia (Investigations) | 6 (6)
Memory impairment (General disorders) | 1 (1)
Muscle weakness (General disorders) | 1 (1)
Pain: Muscle (General disorders) | 4 (5)
Nail changes (General disorders) | 2 (2)
Pain: Extremity-limb (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Palpitations (General disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 2 (2)
International Normalized Ratio of prothrombin time (Investigations) | 1 (1)
Hemorrhage, GI: Rectum (Blood and lymphatic system disorders) | 1 (1)
Pain: Kidney (General disorders) | 1 (1)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 6 (6)
Hyperpigmentation (General disorders) | 1 (1)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 1 (1)
Pain: Urethra (General disorders) | 1 (1)
Hemorrhage Bladder (Vascular disorders) | 1 (1)
Urinary with low grade neutropenia (Infections and infestations) | 1 (1)
Lymphatics - Other (Blood and lymphatic system disorders) | 1 (1)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 7 (7)
Infection with unknown ANC Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal nerve dysfunction (Nervous system disorders) | 1 (1)
Syndromes - Other (General disorders) | 1 (1)
hypocalcemia (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
the worst adverse event of each type was recorded for the course of treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes